CLINICAL TRIAL: NCT04825197
Title: Effects of Late Surfactant Treatment Delivered After a Recruitment Maneuver on Respiratory Outcomes in Extremely Low Gestational Age Newborns: a Randomized Controlled Trial - LATE-REC-SURF Trial
Brief Title: Late Surfactant After a Recruitment Maneuver in Extremely Low Gestational Age Newborns - LATE-REC-SURF Trial
Acronym: LateRecSurf
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: VENTO GIOVANNI (Other)
Responsible Party: Sponsor-Investigator, VENTO GIOVANNI, Associate Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Organization: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3435
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Bronchopulmonary Dysplasia; Chronic Pulmonary Insufficiency of Prematurity
Keywords: surfactant; preterm; recruitment; bronchopulmonary dysplasia; hfov
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth | interventions — poractant alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LRS Group (Experimental): This arm will receive up to 4 doses (100 mg Kg) of Poractant alfa (Curosurf, Chiesi) every 12 hours; each dose preceded by a recruitment manoeuvre in HFOV. Optimal recruitment is defined as adequate oxygenation using a fraction of inspired oxygen (FiO2) of 0.30 or less. The continuous distending pressure (CDP) will be increased stepwise (1 cmH2O every 2-3 min) as long as pulse oximetry (SpO2) improves. The FiO2 will be reduced stepwise, keeping SpO2 within the target range (87-94 %). The recruitment procedure will be stopped if oxygenation no longer improves or if the FiO2 is equal to or less than 0.30. The corresponding CDP will be called the opening pressure (CDPO). Next, the CDP will be reduced stepwise (1-2 cmH2O every 2-3 min) until the SpO2 deteriorates (by at least 2-3 points). The corresponding CDP will be called the closing pressure (CDPC). After a second recruitment maneuver at CDPO for 5 min, the optimal CDP (CDPOPT) will be set 2 cmH2O above the CDPC for at least 3 min.
  Interventions: Drug: Poractant Alfa Intratracheal Suspension [Curosurf]
- Standard Group (No Intervention): This arm will be managed following the ward standard ventilatory protocol which does not contemplate neither surfactant administration nor recruitment manoeuvre.

INTERVENTIONS:
Drug: Poractant Alfa Intratracheal Suspension [Curosurf] — up to 4 doses (100 mg Kg) of Poractant alfa every 12 hours; each dose preceded by a recruitment manoeuvre in HFOV.
  Other Names: Surfactant endotracheal administration following a recruitment HFOV manoeuvre
  Arms: LRS Group

SUMMARY:
This is an unblinded monocentric pilot superiority trial that will be conducted in a IIIlevel NICU at Fondazione Policlinico Agostino Gemelli - IRCCS. The aim of the study is to test the hypothesis that endotracheal administration of poractant alfa preceded by a recruitment manoeuvre in High-Frequency Oscillatory Ventilation (HFOV) modality in preterm infants still requiring mechanical ventilation at 7-10 days of life could reduce the length of invasive mechanical ventilation. Extremely low gestational age newborn infants (GA < 28 weeks) still requiring invasive mechanical ventilation at a postnatal age between 7 and 10 days will be eligible for the study. The study population will be randomly assigned to experimental protocol or to standard care.

Treatment group will receive up to 4 doses (100 mg Kg) of Poractant alfa every 12 hours; each dose will be preceded by a recruitment manoeuvre in HFOV.

Primary endpoint will be the first successful extubation defined as extubation not followed by a reintubation for at least 7 days. Several secondary endpoints will be collected, including respiratory status at one year of age.

DETAILED DESCRIPTION:
Rationale and plausibility of the study. Despite the recent advances in perinatal care, bronchopulmonary dysplasia (BPD) still represents one of the most devastating conditions in premature infants with longstanding consequences on pulmonary function and neurodevelopmental outcomes. Affected infants have a high risk of cerebral palsy and lower cognitive and language skills. Moreover, children with a history of BPD are at a higher risk for developing pulmonary hypertension (PH) and cardiac dysfunction. Despite over 50 years of efforts that have resulted in significant improvements in the care of premature infants, including antenatal glucocorticoid treatment, exogenous surfactant administration, gentler ventilation techniques, judicious use of fluids, prevention of infections and improved nutrition, the incidence of BPD has remained essentially unchanged. BPD is a complex condition that has a multifactorial pathogenesis. Key contributors include oxygen toxicity, ventilator-induced lung injury, inflammation and an arrest of lung vascular development. Multiple animal models and examination of autopsy samples of infants with BPD have confirmed an arrest of vascular development and a simplification of the distal lung architecture as a result of preterm birth and associated lung injury. Indeed, alveolar septation can be preserved in animal models by decreasing the effects of contributors to BPD pathogenesis, including inflammation, oxygen and mechanical ventilation (MV). MV is undoubtedly one of the key advances in neonatal care. Even in this era of noninvasive respiratory support, MV remains a mainstay of therapy in the extremely preterm population. Among survivors, almost 95% of preterm infants were invasively ventilated at some point during their hospital stay. Nevertheless, MV represents one of the major risk factor for BPD. The patient determinants of VILI include preexisting lung injury, lung inflammation and surfactant abnormalities. Premature infants are prone to develop lung atelectasis because of anatomic and functional immaturity of the respiratory system. Further, these infants have lower lung tissue resilience due to deficiency of the following: mature collagen and elastin elements, surfactant and anti-oxidants in their lungs. Therefore, premature infants have a higher incidence of biophysical and biochemical lung injury when subjected to an insult such as mechanical ventilation. In summary, VILI results in an inflammatory cascade that disrupts signaling pathways involved in lung development and repair and contributes to the development of BPD. Therefore, the best strategy to prevent VILI is to avoid mechanical ventilation if possible. Barotrauma, volutrauma, atelectrauma and biotrauma are the major ventilator determinants of VILI. Severe lung inflammation can result in systemic inflammatory response syndrome and multiorgan dysfunction. This pathological process can be mistaken for neonatal sepsis resulting in exposure of these patients to unnecessary antibiotics, which in fact may alter the respiratory microbiome and paradoxically worsen their lung injury. Ventilator-induced lung injury (VILI) represents an ever-present danger for patients in respiratory failure, even in the adult patients. MV can mean irreparable and eventually fatal further damage for the already injured lung. Lung injury is invariably accompanied by alterations in the mechanical properties of the lung itself. There are a variety of microscale structures that contribute to the determination of lung compliance, and that can become altered in acute lung injury. The most severe mechanical consequences of acute lung injury occur when edematous material arising from the vasculature breaches the epithelial barrier and accumulates in the airspaces. Potentially the edematous material interferes with the functioning of pulmonary surfactant in the aerated regions, which is readily accomplished by the plasma proteins via their competition at the air-liquid interface with surfactant. The resulting elevation in surface tension can dramatically reduce compliance and thus the pressure required to ventilate the lung. Elevated surface tension can also prevent inspiratory pressures from prying apart the walls of alveoli and airways that have come into apposition at the end of expiration (atelectasis) or from eliminating plugs of fluid that have formed to occlude small airways. Lung regions that are isolated from ventilation are derecruited. Thus, MV can interfere with surfactant metabolism and function leading to a worse respiratory condition and the need of aggressive ventilation which in turn increases lung injury. The application of mechanical ventilation alone alters surfactant and growth factor expression. Moreover, episodes of increased requirement for ventilatory support are associated with dysfunctional surfactant, which is primarily due to low surfactant protein B (SP-B). Pulmonary surfactant is a complex mixture of phospholipids and proteins that reduce surface tension at the air-liquid interface of the alveolus, thus preventing its collapse during end-exhalation. Surfactant is synthesized and secreted by Type II alveolar epithelial cells, also called pneumocytes, which differentiate between 24 and 34 weeks of gestation in the human. It is made up of 70% to 80% phospholipids, approximately 10% protein and 10% neutral lipids, mainly cholesterol. Surfactant increases surface pressure while lowering surface tension. High surface pressure resists a decrease in alveolar surface area, while low surface tension stabilizes the lung by decreasing the pressure gradient across the alveolar lining layer. Pulmonary surfactant is synthesized, assembled, transported and secreted into the alveolus where it is degraded. It is then recycled in a highly complex and regulated mechanism. This process is slower in newborns (especially those born prematurely) than in adults or those with lung injury. Recently, two randomized controlled trials evaluated the effect of a late surfactant administration in preterm infants with severe respiratory distress that required prolonged invasive ventilation. They failed to demonstrate a reduction in the incidence of BPD at 36 wks postmenstrual age (PMA) among infants treated with late surfactant but showed some improvements in long-terms outcomes (less rehospitalization for pulmonary problems and less use of home respiratory support over the first year of life) (9-10). Moreover, in the study by Hascoet et al, the 2-year follow-up showed a statistically significant better growth among the treatment group patients compared to the control group ones. Nevertheless, both the studies were designed in order to show an improvement in short-term outcomes as the day of the first successful extubation or the BPD rate, but in nor in the first study neither in the former one they achieved the hoped results. Indeed, the above-mentioned trials were inconclusive but encouraging, as they failed to demonstrate the objective they were designed for but still showed some good results in terms of long-term outcomes (respiratory morbidity at one year of age and growth at two years of age). As well as the ineffective results, there are some differences in the study design among the two trials that weaken the conclusion of both the trials. In the study by Hascoet et al, a single dose of 200mg/kg of poractant alfa was administered at 14 days of life. In the TOLSURF study, patients were randomized between 7 and 14 days of life and received up to 5 doses of calfactant associated to iNO therapy. In neither of the two trials surfactant was preceded by a recruitment manoeuvre. In animal models, lung recruitment before surfactant administration improved gas exchange and lung function owing to a more homogeneous surfactant distribution. We hypothesized that optimizing end-expiratory lung volume before surfactant administration may improve the success rate of a late treatment with surfactant.

Safety. Based on the available literature regarding the recruitment maneuver and the administration of Curosurf in premature infants, it is reasonable to expect from the treatment an improvement in respiratory conditions and consequently an earlier extubation of the treated infants, that would lead to several beneficial consequences on respiratory and neurological outcomes in the medium and long term. At the same time, the risk associated with the procedure is the occurrence of the most common side effects of the procedure and the drug in this subsets of premature newborns (ELGANS at 10 days of life): hemodynamically significant PDA that requires pharmacological treatment or pneumothorax that requires chest drainage. Since they are both common pathological conditions in premature infants, there are available safe treatments in neonatal intensive care units. Safety will be evaluated daily during the treatment period. An additional safety evaluation will be performed at discharge and at the final study visit (follow up visit).

Monitoring. The trial will be conducted in accordance with the current approved protocol, ICH GCP, relevant regulations, and standard operating procedures. The Sponsor's designees will monitor all aspects of the study carefully with respect to ICH GCPs and SOPs for compliance with applicable government regulations. The investigator is responsible for providing all study records, including eCRFs, source documents, etc., for review and inspection by the clinical monitor. eCRF will be periodically monitored and source verified against corresponding source documentation (e.g., office and clinical laboratory records) for each subject. Clinical monitors will evaluate periodically the progress of the study, including the verification of appropriate consent form procedures, review of drug accountability and study drug preparation procedures, adherence to dosing procedures, the investigator's adherence to the protocol, maintenance of records and reports, review of source documents for accuracy, completeness, and legibility, and review of study regulatory documents, including, but not limited to: study agreement, study insurance. Moreover, monitoring activities will be also conducted by an external society, independent from the sponsor. In addition, the monitor shall review completed eCRF and study documentation for accuracy and completeness, and protocol compliance. The monitor will assure that data captured in the eCRF is fully supported by the source documents.

End of the study. This study will end when the last patient randomized will be visited at one year of age for the last follow-up visit.

Randomisation. Infants will be allocated to one of the two groups in the ratio 1:1 according to the minimization method. Following screening procedures eligible infants will be randomly assigned to one of the two treatment groups. Randomization will be performed using random allocation generated by computer code. The randomization will be performed in permuted unequal blocks. The random allocation sequence will be generated using the module ralloc.ado in Stata/IC 16.1 (Stata-Corp, College Station, Texas). Concealment will be performed by closed envelopes.

Statistics. No formal sample size calculation was performed because this is a pilot study. Revising our past records, we estimate that there will be a number of 20-25 patients having the eligibility criteria in the study period. Therefore, we chose to recruit 10 patients in each group. Clinical characteristics of infants will be described using mean values and standard deviation, median value and range, or rate and percentage. Univariate statistical analysis will be performed using the Student "t" test for parametric continuous variables, the Wilcoxon rank-sum test for non-parametric continuous variables, and Fisher's exact test for categorical variables. A p <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 1. Extremely low gestational age newborn infants (GA < 28 weeks) - gestational age matching between maternal dates and/or early antenatal ultrasound
* 2. Singleton or multiple birth
* 3. Postnatal age between 7 and 10 days
* 4. Invasive mechanical ventilation still needed
* 5. Fraction of inspired oxygen (FiO2) of more than 0.30 and/or an oxygenation index of 8 or more for at least 6 hours
* 6. Stable cardiovascular condition
* 7. Informed consent form signed by parents or legal guardian

Exclusion Criteria:

* 1. Major congenital malformation (i.e., infants with genetic, metabolic or endocrine disorder diagnosed before enrolment)
* 2. High index of suspicion of infection before enrolment
* 3. Neurological conditions that might contraindicate extubation
* 4. Inotropic agents needed
* 5. Pneumothorax
* 6. Hemodynamically significant ductus arteriosus
* 7. Surgical intervention within the past 72 hours
* 8. Partecipation in another interventional clinical study that may interfere with the results of this trial
* 9. Known hypersensitivity to the drug or to one of the excipients

Ages: 7 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
First successful extubation | From date of randomization until the date of first documented progression, assessed up to 40 weeks of post menstrual age
  The time to first successful extubation ( expressed as day of life).

SECONDARY OUTCOMES:
Rate of Bronchopulmonary dysplasia | At 36 weeks of post-menstrual age
  Oxygen-dependance at 36 weeks of post-menstrual age
Rate of Interstitial emphysema | In the 21 days following experimental treatment
  Xray-documented
Rate of Pneumothorax | In the 21 days following experimental treatment
  Ultrasound or Xray-documented
Rate of Pulmonary haemorrhage | In the 21 days following experimental treatment
  Clinically diagnosed
Rate of Necrotising enterocolitis | Up to 40 weeks post-mestrual age
  Bell's Criteria
Rate of intraventricular haemorrhage | From date of randomization - up to 40 weeks post-mestrual age
  Ultrasound documented intraventricular haemorrhage of any grade (Volpe's classification)
Rate of Periventricular leukomalacia | From date of randomization up to 40 weeks post-mestrual age
  Ultrasound documented periventricular leukomalacia (DeVries's classification)
Length of hospital stay | Through study completion, an average of 1 year
  Number of days of hospital stay
Length of invasive mechanical ventilation | Up to 40 weeks post-mestrual age
  Number of days of invasive mechanical ventilation
Length of oxygen-therapy | Up to 40 weeks post-mestrual age
  Number of days of oxygen-therapy
Length of respiratory support | Up to 40 weeks post-mestrual age
  Number of days of respiratory support
Use of postnatal steroids | Up to 40 weeks post-mestrual age
  Use of postnatal steroids to prevent or treat bronchopulmonary dysplasia
Rehospitalisation for respiratory problems in the first year of life | One year of life
  Number of rehospitalisation for respiratory problems in the first year of life

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Vento, Professor, Principal Investigator — Fondazione Policlinico Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 6 months following article publication.
Access Criteria: All researchers who provide a methodologically sound proposal will have access to data. Proposals should be directed to giovanni.vento@unicatt.it.

REFERENCES:
- [Background] Bates JHT, Smith BJ. Ventilator-induced lung injury and lung mechanics. Ann Transl Med. 2018 Oct;6(19):378. doi: 10.21037/atm.2018.06.29. PMID 30460252
- [Background] Digeronimo RJ, Mustafa SB, Ryan RM, Sternberg ZZ, Ashton DJ, Seidner SR. Mechanical ventilation down-regulates surfactant protein A and keratinocyte growth factor expression in premature rabbits. Pediatr Res. 2007 Sep;62(3):277-82. doi: 10.1203/PDR.0b013e3181256aeb. PMID 17622950
- [Background] Merrill JD, Ballard RA, Cnaan A, Hibbs AM, Godinez RI, Godinez MH, Truog WE, Ballard PL. Dysfunction of pulmonary surfactant in chronically ventilated premature infants. Pediatr Res. 2004 Dec;56(6):918-26. doi: 10.1203/01.PDR.0000145565.45490.D9. Epub 2004 Oct 20. PMID 15496605
- [Background] Hascoet JM, Picaud JC, Ligi I, Blanc T, Moreau F, Pinturier MF, Zupan V, Guilhoto I, Hamon IR, Alexandre C, Bouissou A, Storme L, Patkai J, Pomedio M, Rouabah M, Coletto L, Vieux R. Late Surfactant Administration in Very Preterm Neonates With Prolonged Respiratory Distress and Pulmonary Outcome at 1 Year of Age: A Randomized Clinical Trial. JAMA Pediatr. 2016 Apr;170(4):365-72. doi: 10.1001/jamapediatrics.2015.4617. PMID 26928567
- [Background] Ballard RA, Keller RL, Black DM, Ballard PL, Merrill JD, Eichenwald EC, Truog WE, Mammel MC, Steinhorn RH, Rogers EE, Ryan RM, Durand DJ, Asselin JM, Bendel CM, Bendel-Stenzel EM, Courtney SE, Dhanireddy R, Hudak ML, Koch FR, Mayock DE, McKay VJ, O'Shea TM, Porta NF, Wadhawan R, Palermo L; TOLSURF Study Group. Randomized Trial of Late Surfactant Treatment in Ventilated Preterm Infants Receiving Inhaled Nitric Oxide. J Pediatr. 2016 Jan;168:23-29.e4. doi: 10.1016/j.jpeds.2015.09.031. Epub 2015 Oct 21. PMID 26500107
- [Background] Tingay DG, Togo A, Pereira-Fantini PM, Miedema M, McCall KE, Perkins EJ, Thomson J, Dowse G, Sourial M, Dellaca RL, Davis PG, Dargaville PA. Aeration strategy at birth influences the physiological response to surfactant in preterm lambs. Arch Dis Child Fetal Neonatal Ed. 2019 Nov;104(6):F587-F593. doi: 10.1136/archdischild-2018-316240. Epub 2019 Feb 1. PMID 31498776
- [Background] Vento G, Ventura ML, Pastorino R, van Kaam AH, Carnielli V, Cools F, Dani C, Mosca F, Polglase G, Tagliabue P, Boni L, Cota F, Tana M, Tirone C, Aurilia C, Lio A, Costa S, D'Andrea V, Lucente M, Nigro G, Giordano L, Roma V, Villani PE, Fusco FP, Fasolato V, Colnaghi MR, Matassa PG, Vendettuoli V, Poggi C, Del Vecchio A, Petrillo F, Betta P, Mattia C, Garani G, Solinas A, Gitto E, Salvo V, Gargano G, Balestri E, Sandri F, Mescoli G, Martinelli S, Ilardi L, Ciarmoli E, Di Fabio S, Maranella E, Grassia C, Ausanio G, Rossi V, Motta A, Tina LG, Maiolo K, Nobile S, Messner H, Staffler A, Ferrero F, Stasi I, Pieragostini L, Mondello I, Haass C, Consigli C, Vedovato S, Grison A, Maffei G, Presta G, Perniola R, Vitaliti M, Re MP, De Curtis M, Cardilli V, Lago P, Tormena F, Orfeo L, Gizzi C, Massenzi L, Gazzolo D, Strozzi MCM, Bottino R, Pontiggia F, Berardi A, Guidotti I, Cacace C, Meli V, Quartulli L, Scorrano A, Casati A, Grappone L, Pillow JJ. Lung recruitment before surfactant administration in extremely preterm neonates with respiratory distress syndrome (IN-REC-SUR-E): a randomised, unblinded, controlled trial. Lancet Respir Med. 2021 Feb;9(2):159-166. doi: 10.1016/S2213-2600(20)30179-X. Epub 2020 Jul 17. PMID 32687801
- [Background] Shalish W, Kanbar L, Keszler M, Chawla S, Kovacs L, Rao S, Panaitescu BA, Laliberte A, Precup D, Brown K, Kearney RE, Sant'Anna GM. Patterns of reintubation in extremely preterm infants: a longitudinal cohort study. Pediatr Res. 2018 May;83(5):969-975. doi: 10.1038/pr.2017.330. Epub 2018 Jan 31. PMID 29389921